CLINICAL TRIAL: NCT03884127
Title: Analysis of Changes in Intestinal Flora of Hyperlipidemia by Ezetimibe and Orlistat.
Brief Title: Ezetimibe and Orlistat Affect the Intestinal Flora of Hyperlipidemia.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fifth Affiliated Hospital of Xinjiang Medical University (Other)
Collaborators: West China Hospital (Other)
Responsible Party: Principal Investigator, Jin jin, physician, Fifth Affiliated Hospital of Xinjiang Medical University
Other Study IDs: FifthXinjiang
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-02

CONDITIONS: Hyperlipidemia
Keywords: orlistat; Ezetimibe; Gastrointestinal Microbiome
MeSH Terms: conditions — Hyperlipidemias | interventions — Ezetimibe; Orlistat

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal bacteria DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- hyperlipidaemia: On the basis of the intervention of therapeutic sexual life style, a case control study was conducted on the intervention of oral ezetimibe tablet and orlistat capsule for 12 weeks and hyperlipidemia patients who persisted in the use of basic treatment.
  Interventions: Drug: Ezetimibe 10mg; Drug: Orlistat 120 MG

INTERVENTIONS:
Drug: Ezetimibe 10mg — On the basis of the intervention of life style, drug intervention therapy was carried out for a period of 12 weeks
  Other Names: lifestyle intervention
Drug: Orlistat 120 MG — On the basis of the intervention of life style, drug intervention therapy was carried out for a period of 12 weeks
  Other Names: lifestyle intervention

SUMMARY:
At present,the prevalence of hyperlipidemia in Chinese adults is 40.40%,which is related to atherosclerotic cardiovascular disease and diabetes independent risk factors,while increasing the risk of cancer.Lipid metabolism affects the nutritional status of the intestinal epithelium,making the intestine Changes in the microenvironment of the intestinal flora affect the distribution of intestinal flora and eventually lead to bile acid metabolism change.Bile acid is a signal molecule that regulates glucose and lipid and energy metabolism in vivo State.The regulation of intestinal flora may be a new way to treat the imbalance of lipid metabolism,but it is currently sensitive to lipid metabolism the microbiome studies are unclear.In this study, newly diagnosed overweight patients with hyperlipidemia were treated with cholesterol absorption inhibition The drug intervention of ezeomab tablet and orlistat capsule for 12 weeks was observed to observe the changes of intestinal flora and bile acid metabolism after excessive cholesterol and triglyceride production.Clinical screening for the treatment of hyperlipidemia the study provides a reference for bacteria species and prevention and treatment,and provides a research basis for further development of drugs or foods that interfere with lipid metabolism by interfering with intestinal flora.

DETAILED DESCRIPTION:
1. Research background;Currently, hyperlipidemia in Chinese adults is 40.40%, and is an independent risk factor for atherosclerotic cardiovascular disease and diabetes, as well as increasing the risk of tumor.Hyperlipidemia and intestinal flora are closely related and interact with each other. Intervention of intestinal flora may be one of the ways to treat hyperlipidemia.
2. Research objective: to observe the changes of intestinal flora in obese patients with hyperlipidemia who have indications of lipase absorption inhibitor orlistat and cholesterol absorption inhibitor ezeomab and analyze the related influencing factors.
3. Research methods and procedures; 3.1 on the basis of community people, on the basis of the baseline survey, choosing a new diagnosis of overweight patients with hyperlipidemia, to carry out the treatment of sexual lifestyle intervention therapy on the basis of oral respectively in accordance with the wheat cloth folding, orlistat capsules for 12 weeks intervention and consistent use of foundation treatment in patients with hyperlipidemia and case-control study.

3.2 on the basis of the indications and voluntary choice of newly diagnosed patients with hyperlipidemia, overweight in the treatment of sexual lifestyle intervention therapy on the basis of, to carry out the drug intervention therapy for 12 weeks, oral respectively according to the fold of wheat and cloth (10 mg, 1 time/day), orlistat capsules (120 mg, 2-3 times/day) to intervene with consistent use of foundation treatment in patients with hyperlipidemia control study.

3.3 telephone follow-up and outpatient follow-up were adopted.All subjects were closely followed up to observe the changes of the patient's condition and whether there were adverse reactions.At the end of 12 weeks of the experiment, blood was drawn on an empty stomach in the morning, and fasting was started after dinner the day before the experiment. The duration of fasting was not less than 8-10 hours, and drinking water was allowed.Three blood samples were collected.

3.4 experiment for the first time in the morning on the day of gathering patients out of fresh 10 g, solid manure into the sterile collection box of oil fecal DNA protection (liquid), the stool specimens in the laboratory is divided into four, then immediately put - 80 ℃ low temperature refrigerator or liquid nitrogen preservation, stay late in intestinal flora DNA extraction.real 4, participants accept blood fat, this is one of the clinical routine physical examination project, orlistat capsules of non-prescription drugs is losing weight, but the existing studies show that after the application of the drug can bring benefit of blood sugar, blood lipid, body weight, and in accordance with the folding mab are clinical commonly used drugs, both has the effect of reducing blood fat, reducing blood fat, bring to significant cardiovascular benefits, and compared with statins, there is no evidence that these drugs can increase the risk of new diabetes.

Subjects can learn about their health conditions in terms of blood lipids through testing. The relevant information obtained from subjects can be used for clinical diagnosis and treatment of hyperlipidemia and contribute to the prevention and treatment of hyperlipidemia.In this study, relevant samples were stored in the endocrine and metabolic diseases laboratory of west China hospital.The researcher promises that the samples will only be used for this study, and will not disclose the samples, patients' clinical information and other data to irrelevant personnel in this study.Clinical data collection (demographic data, measured blood pressure, height, weight, etc.), blood lipids, and intestinal flora monitoring were all undertaken by researchers.The registration fee incurred on the day of inspection shall be borne by the researcher, and the meal fee and transportation fee incurred on the day shall be subsidized to a certain extent (RMB fifty). The financial burden of the subject will not be increased during the whole experiment.

5. Alternative methods of diagnosis and treatment. According to the 2016 Chinese adult guidelines for the prevention and treatment of dysmatosis in Chinese adults (revised version in 2016), subjects may choose other kinds of appropriate drugs, such as statins, betins, niacin, bile acid chelating agents, etc., at their own expense.

ELIGIBILITY:
Inclusion Criteria:

(1) according to the guidelines for the prevention and treatment of dyslipidemia in Chinese adults (revised in 2016), the diagnostic criteria for hyperlipidemia were met, and the stratification criteria for dyslipidemia in Chinese ASCVD primary prevention population were: TC greater than or equal to 6.2mmol/l, ldl-c greater than or equal to 4.1mmol/l, non-hdl-c greater than or equal to 4.9mmol/l, and TG greater than or equal to 2.3mmol/l.(2) newly diagnosed hyperlipidemia patients, BMI 24kg/m2, did not take any lipid-regulating or lipid-lowering drugs within a month;(3) exclude obvious cardiovascular and cerebrovascular diseases by medical history inquiry, physical examination, electrocardiogram examination, skull imaging examination and other data;(4) mental health, after informed consent to participate in the study.

Exclusion Criteria:

(1)acute and chronic liver, renal insufficiency, cholestasis;Acute infectious diseases;Malignant tumor;Thyroid disease;Diseases of the immune system;Patients with gastrointestinal diseases;(2)patients with severe mental illness and cognitive impairment;(3) have used the drugs that have an impact on this study before treatment;(4)allergic to the study of drugs, drug side effects can not be tolerated, do not want to take biological specimens;(5)pregnant and nursing women;6. Did not sign the informed agreement;(7)the use of antibiotics, probiotics and other drugs to interfere with intestinal flora, health products, etc.,in the last 3 months.All experiments were conducted in accordance with relevant legal and institutional guidelines.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: On the basis of the community population, the newly diagnosed overweight and hyperlipidemia patients were selected on the basis of baseline investigation
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
blood lipid | enroll(0 month)，finish(3 month)
  Triglycerides, total cholesterol, LDL cholesterol, HDL cholesterol
bile acid | enroll(0 month)，finish(3 month)
  total bile acid
Gastrointestinal flora | enroll(0 month)，finish(3 month)
  Firmicutes, bacteroides

CONTACTS AND LOCATIONS:
Overall Officials: haoming tian, master, Study Chair — West China Hospital

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed, the results will be uploaded
Supporting Information: Study Protocol, CSR
Time Frame: starting 6 months after publication
Access Criteria: In excel form,include Baseline data, post-intervention outcomes